CLINICAL TRIAL: NCT00445549
Title: Phase II Study of Clinical Activity and Proteomic Pathway Profiling of the Vascular Endothelial Growth Factor 2 (VEGFR2) Inhibitor, ZD6474 (Vandetanib) in Women With Relapsed or Refractory Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Vandetanib to Treat Women With Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study closed because of inadequate early activity.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Elise C. Kohn, M.D., National Cancer Institute (NCI), National Institutes of Health (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070061; 07-C-0061 (Other: Clinical Center (CC), National Institutes of Health (NIH)); 070061 (Other: Clinical Center (CC), National Institutes of Health (NIH))
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-05

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms
Keywords: Ovarian; VEGFR2; EGFR; Angiogenesis; Tyrosine Kinase; Protein Phosphorylation; Vandetanib; Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vandetanib treatment (Experimental): 300 mg daily oral dose, 28 day cycle
  Interventions: Drug: Vandetanib

INTERVENTIONS:
Drug: Vandetanib — 300 mg daily dose, 28 day cycle
  Other Names: Zactima; ZD6474

SUMMARY:
Background:

* Vandetanib is a drug that attacks a group of proteins on the surface of many cells, especially blood vessel cells and tumor cells.
* Tumors require the development of new blood vessels in order to grow and spread.
* In laboratory experiments, vandetanib slowed the growth of certain tumors and regulated their blood vessel growth.
* In early clinical trials, some patients' tumors did not grow for a period of time while they were receiving vandetanib.

Objectives:

* To determine whether vandetanib can cause tumors to shrink or stabilize in some patients with ovarian cancer, fallopian tube cancer or primary peritoneal cancer.
* To determine, by tumor biopsy, if features of the tumor change with vandetanib treatment may predict if the tumor will likely respond to vandetanib.

Eligibility:

* Women 18 years of age and older with ovarian, fallopian tube or primary peritoneal cancer that does not respond to standard treatment.

Design:

* Patients take vandetanib daily, by mouth in 28-day cycles until their disease worsens or they develop unacceptable side effects.
* Tumor biopsies (surgical removal of a sample of tumor tissue) are done before starting vandetanib treatment and after 6 weeks of treatment.
* Patients are followed in the clinic every 4 weeks during treatment for a physical examination, blood tests, and review of laboratory studies and side effects.
* Patients have a computed tomography (CT) scan every 8 weeks to monitor tumor growth and magnetic resonance imaging (MRI) before starting vandetanib treatment, on the third day after taking vandetanib and 6 weeks into treatment.
* Patients quality of life is assessed with regularly scheduled questionnaires.

DETAILED DESCRIPTION:
Background:

* Epithelial ovarian cancer requires neovascularization for growth and metastasis. Anti-angiogenesis agents have been shown to have promise in the treatment of recurrent disease. Expression of vascular endothelial growth factor 2 (VEGFR2) and epidermal growth factor receptor (EGFR) has been demonstrated in ovarian cancer specimens in stroma and tumor. Blocking autocrine and paracrine loops acting through these receptors may inhibit downstream phosphorylation targets in the mitogen activated protein kinase (MAPK) and AKT pathways, thereby influencing disease progression and patient outcome.
* The multi-kinase inhibitor ZD6474 (vandetanib, AstraZeneca, Zactima) blocks angiogenesis by targeting VEGFR2, and shows in vitro activity against a number of other receptor tyrosine kinases including resonance energy transfer (RET), vascular endothelial growth factor 3 (VEGFR3) and EGFR.
* Clinical efficacy of ZD6474 (vandetanib) in women with refractory or relapsed epithelial ovarian cancer is unknown, but preclinical data suggests potential value.
* The maximum tolerated dose of ZD6474 (vandetanib) has been determined at 300mg/day, limited by the dose-responsive adverse effect of prolonged (Q wave, T wave)QT interval.

Objectives:

* To assess the clinical activity (CR - complete response, PR - partial response, or disease stabilization) of the VEGFR2 inhibitor ZD6474 (vandetanib), 300mg/d, in women with ovarian, fallopian tube or primary peritoneal cancer.
* To study target signal events: quantity and activation of VEGFR2, EGFR, AKT and extracellular signal-regulated kinases (ERK).

Eligibility:

* Women with biopsy-proven epithelial ovarian, fallopian tube or primary peritoneal cancer that is relapsed and/or refractory to prior therapy.
* Women must have measurable disease by NCI Response Evaluation Criteria in Solid Tumors (RECIST) criteria and a sentinel lesion adequate for core biopsy through percutaneous biopsy.
* Women must have had no more than four prior treatment regimens.

Design:

* Women will receive 300mg of ZD6474 (vandetanib) daily, orally in 28-day cycles until disease progression, excessive toxicity, or withdrawal from study.
* Biopsy of tumor will be performed prior to starting ZD6474 (vandetanib) and after six weeks of treatment. The quantity of phosphorylated VEGFR2, EGFR, ERK and AKT in the biopsy tissue will be analyzed.
* Clinical outcome and toxicity will be measured and correlated with target inhibition.
* Women will also undergo serial imaging with dynamic contrast-enhanced MRI to estimate tumor blood flow.
* Research blood samples will be taken to assess changes in circulating cytokine concentrations.
* Quality of life will be assessed during treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years and older with biopsy-proven epithelial ovarian, fallopian tube or primary peritoneal cancer that is relapsed or refractory to prior standard platinum-and taxane based therapy will be eligible.
* Histopathologic diagnosis must be confirmed in the Laboratory of Pathology (LP), NCI. A block of the primary or later access to recut slides is required. If this is unavailable, a recent resection of a metastatic site is required for entry.
* All patients must have measurable disease by NCI RECIST criteria and a sentinel lesion adequate for core biopsy through percutaneous biopsy.
* Patients must have a performance status of Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2.
* Patients must have good end organ function:
* white blood cells (WBC) greater than 3000/mm(3)
* absolute neutrophil count (ANC) greater than 1000/mm(3)
* platelets greater than 150,000/mm(3)
* serum creatinine less than 1.5 mg/dl
* liver function tests (AST and ALT) within 2.5 times the upper limit of normal (ULN)
* bilirubin less than 1.5 mg/dl
* potassium between 4.0 and ULN (supplementation allowed)
* magnesium (Mg) and calcium (Ca) within normal limits (supplementation allowed)
* Systolic blood pressure less than 160 mm Hg and diastolic blood pressure less than 100 mm Hg (therapy permitted)
* Patients must be at least 4 weeks from previous therapy (chemotherapy, hormonal therapy, and radiation therapy, alternative therapy or investigational agents). Carboplatin, must not have been received for at least 6 weeks prior to enrollment.
* Patients must have received no more than 4 prior regimens for the treatment of ovarian cancer.
* Patients must have recovered from any toxicity related to prior cancer therapy to NCI grade 1, except for peripheral neuropathy, which must have recovered to grade 2 or better.
* Women of childbearing age and potential must agree to use adequate barrier contraception (interaction with oral contraceptives is unknown) prior to study entry, during therapy and for 3 months after completion of therapy.
* Patients must be able to give written informed consent.
* All eligible patients must be registered by contacting Central Registration personnel by fax at (301) 480-0757 between the hours of 8:30am and 5:00 pm, Monday through Friday.

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigators opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Evidence of central nervous system (CNS) involvement (patients with abnormal clinical exam or history will require a head CT or MRI.
* History of cardiac disorders including:
* Clinically significant cardiac event such as myocardial infarction, New York Heart Association (NYHA) classification of heart disease greater than or equal to 2 within 3 months of entry, or presence of cardiac disease that, in the opinion of the investigator,increases the risk of ventricular arrhythmia.
* Uncontrolled arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic.
* Previous history of medication-induced corrected QT interval (QTc) prolongation requiring discontinuation of that medication.
* Congenital long (Q wave, T wave) QT syndrome, or 1st degree relative with unexplained early sudden cardiac death(less than 40 years of age).
* Presence of left bundle branch block (LBBB).
* QTc, corrected per automated electrocardiogram (ECG) standards, that is unmeasurable, or greater than or equal to 480 msec on screening ECG. If a patient has QTc greater than or equal to 480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be less than 480 msec in order for the patient to be eligible for the study.
* Patients requiring any concomitant treatment with medication that may cause QTc prolongation or induce Torsades de Pointes will not be permitted to enter this study unless the agent can safely be changed to one not affecting QTc.
* Patients requiring any concomitant treatment with medication that may inhibit (cytochrome p450 3A4) CYP3A4 will not be permitted to begin this study. If it is considered medically safe to discontinue such medication, the patient may become eligible once a sufficient amount of time after the last dose of such medications has elapsed to consider the drug adequately eliminated (at least 5 half lives of the drug).
* Patients with active infection will not be eligible, but may become eligible once infection has resolved and they are at least 7 days from completion of antibiotics.
* Patients with incomplete wound healing from previous surgery or injury will be ineligible. Patients must be at least 4 weeks from a major surgical procedure.
* Women who are actively breast-feeding will be excluded.
* Currently active diarrhea that is uncontrolled with medication (e.g. bulk agents or loperamide) that may affect the ability of the patient to absorb the ZD6474.
* Previous or current malignancies within the last 5 years, with the exception of cervical carcinoma in situ curatively treated, ductal or lobular carcinoma in situ curatively treated and without ongoing therapeutic intervention.
* No concomitant use of complementary or alternative medication or other agents (investigational or anti-cancer agents) will be allowed without approval of a principal investigator (PI) or associate investigator (AI). Every effort will be made to maximize patient safety and minimize changes in chronic medications.
* Patients with a history of deep venous thrombosis or pulmonary embolism within the past 3 months or those patients requiring ongoing anticoagulation will be ineligible.
* Patients with a history of gastrointestinal (GI) bleed or gross hematuria within the past 30 days will be ineligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elise C Kohn, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hollingsworth HC, Kohn EC, Steinberg SM, Rothenberg ML, Merino MJ. Tumor angiogenesis in advanced stage ovarian carcinoma. Am J Pathol. 1995 Jul;147(1):33-41. PMID 7541612
- [Background] Spentzos D, Levine DA, Ramoni MF, Joseph M, Gu X, Boyd J, Libermann TA, Cannistra SA. Gene expression signature with independent prognostic significance in epithelial ovarian cancer. J Clin Oncol. 2004 Dec 1;22(23):4700-10. doi: 10.1200/JCO.2004.04.070. Epub 2004 Oct 25. PMID 15505275
- [Background] Ryan AJ, Wedge SR. ZD6474--a novel inhibitor of VEGFR and EGFR tyrosine kinase activity. Br J Cancer. 2005 Jun;92 Suppl 1(Suppl 1):S6-13. doi: 10.1038/sj.bjc.6602603. PMID 15928657
- [Result] Annunziata CM, Walker AJ, Minasian L, Yu M, Kotz H, Wood BJ, Calvo K, Choyke P, Kimm D, Steinberg SM, Kohn EC. Vandetanib, designed to inhibit VEGFR2 and EGFR signaling, had no clinical activity as monotherapy for recurrent ovarian cancer and no detectable modulation of VEGFR2. Clin Cancer Res. 2010 Jan 15;16(2):664-72. doi: 10.1158/1078-0432.CCR-09-2308. Epub 2010 Jan 12. PMID 20068097
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: RECIST — http://ctep.cancer.gov/protocolDevelopment/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: If 2-3 patients per month enroll onto this trial, it is expected that approximately one and a half years will be required to enroll the 35 evaluable patients required for evaluation in this study. To make an allowance for a small drop-out of patients from the study and still preserve the intended accrual goal, the total accrual will be38 patients.
Period: Overall Study
Arm/Group | Vandetanib Treatment
Started | 12
Completed | 0
Not Completed | 12
Not completed — progressive disease | 12

BASELINE CHARACTERISTICS:
Arm/Group | Vandetanib Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 59.13 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Efficacy
Description: Defined as complete response (CR), partial response (PR), or disease stabilization lasting 6 months or longer per RECIST criteria. CR-total disappearance of all evaluable disease. PR->30% reduction in the sum of the longest diameters (LD) of target lesions. Stable disease (SD) is <30% decrease and <20% increase in the sum of the LD of all target lesions. See the protocol Link module for full RECIST criteria.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Vandetanib Treatment
Number analyzed (Participants) | 12
participants | 0 [1 to 6]

2. Secondary Outcome: The Number of Participants With Adverse Events
Description: Here are the total # of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: 22 months
Measure: Number; unit: Participants
Arm/Group | Vandetanib Treatment
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: 22 months
Arm/Group | Vandetanib Treatment
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vandetanib Treatment (N=12)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 8 (15)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 11 (16)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 9 (14)
Alkaline phosphatase (Investigations) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 3 (8)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine (Investigations) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 10 (21)
Distension/bloating, abdominal (Gastrointestinal disorders) | 2 (2)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Edema: limb (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (6)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (3)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (6)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Investigations) | 2 (2)
Hemoglobinuria (Investigations) | 3 (3)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU::Ureter (Renal and urinary disorders) | 1 (1)
Hemorrhage, GU::Vagina (Reproductive system and breast disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes/flushes (Vascular disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vulva (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Vagina (Infections and infestations) | 1 (1)
Infection with unknown ANC::Urinary tract NOS (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (3)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6 (12)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (2)
Obstruction, GI::Small bowel NOS (Gastrointestinal disorders) | 1 (1)
Obstruction, GU::Ureter (Renal and urinary disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Investigations) | 2 (2)
Pain::Abdomen NOS (General disorders) | 5 (6)
Pain::Chest/thorax NOS (General disorders) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 1 (1)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain::Pelvis (Reproductive system and breast disorders) | 1 (1)
Photosensitivity (Eye disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (4)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4 (5)
Prolonged QTc interval (Investigations) | 8 (13)
Proteinuria (Renal and urinary disorders) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6 (8)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 (7)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 4 (5)
Taste alteration (dysgeusia) (Nervous system disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 5 (6)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Weight loss (Investigations) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The study closed after the first stage of accrual because of inadequate early activity with 32 cycles of administered treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No